CLINICAL TRIAL: NCT04019665
Title: Self-screening of Cognitive Impairment in Primary Care: a Comparative Study Between a Test Based on SAGE at Home and MMSE at Doctor's Office in Picardie
Brief Title: Self-screening of Cognitive Impairment in Primary Care
Acronym: OCEANE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2018_843_0024
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Cognition Disorder; Alzheimer Disease
Keywords: Cognition Disorder; Alzheimer Disease; MMSE; SAGE
MeSH Terms: conditions — Cognition Disorders; Alzheimer Disease | interventions — Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAGE and MMSE score (Other)
  Interventions: Other: MMSE (mini mental state examination); Other: SAGE (Self-Administered Gerocognitive Exam)

INTERVENTIONS:
Other: MMSE (mini mental state examination) — mini mental state examination takes place during the consultation. The consultation is a general or post-emergency geriatric consultation.
Other: SAGE (Self-Administered Gerocognitive Exam) — SAGE test contains a series of questions that assess the cognitive functioning. Sage was developed by the Ohio State University Wexner Medical Center. it's an online, at-home, self-screening dementia tool that has been scientifically evaluated, and it's demonstrated good results in accurately identifying cognitive deficits.

SUMMARY:
According to 2011 HAS recommendations, early detection of Alzheimer disease is the major objective in order to allow an earlier care and support. These recommendations strengthen general practitioner role, who plays a key role in the identification of cognitively impaired patients. HAS recommendations are the use of MMSE like test (Mini Mental State Examination) at general practitioner office. A self-screening test, without medical presence, would allow a self-administered cognitive assessment by the patient. A review of the literature about self-administered cognitive tests has been realized. The Self-Administered Gerocognitive Examination (SAGE) has been chosen. It is a brief, valid and reliable cognitive assessment tool, rated on 22 points, which allows an early detection of cognitive impairment, with a sensitivity close to the MMSE test. Nevertheless, SAGE has never been tested at home without medical supervision. In this study, the investigators will determine if SAGE scores at home correlates with MMSE scores at general practitioner office.

Patients with inclusion criteria will be recruited during the general practitioner consultation and will have a clinical assessment included MMSE and clinical data collection. Then, SAGE will be given to the patient in order to be completed at home without medical supervision and send to the general practitioner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects from three Picard general practitioner's practice
* 60 years old or more
* patients who accept to complete the tests
* with ou without cognitive complaint
* patients able to read and write
* affiliated to social security system

Exclusion Criteria:

* major visual disorders
* legal safeguard
* diagnosis of neuro-cognitive disorder

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
MMSE Score at general or post emergency geriatric consultation | day 0
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment.
Sage test done at home | 10 days
  SAGE (Self-Administered Gerocognitive Exam) test, and was developed by the Ohio State University Wexner Medical Center. Average time to complete the test is 15 minutes. The maximum score is 22. A score of 17 and above is considered normal.
Concordance between the MMSE test score done at consultation and the sage test core done at home | 10 days
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. SAGE (Self-Administered Gerocognitive Exam) test, and was developed by the Ohio State University Wexner Medical Center. Average time to complete the test is 15 minutes. The maximum score is 22. A score of 17 and above is considered normal.

CONTACTS AND LOCATIONS:
Overall Officials: Federspiel, MD, Principal Investigator — CHU Amiens; Deschamps, MD, Principal Investigator — Montdidier; Briat-Lagache, MD, Principal Investigator — Hangest-en-Santerre
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No